CLINICAL TRIAL: NCT05101421
Title: The Effects of Rice Ceramide Supplementation in Improving Skin Health
Brief Title: Rice Ceramide Supplementation and Skin Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nexus Wise Sdn Bhd (Industry)
Collaborators: JScience Consultancy PLT (Unknown)
Responsible Party: Principal Investigator, Tan Chung Keat, Clinical Assistant Professor, Nexus Wise Sdn Bhd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NW-RC-001
Record Dates: First submitted 2021-10-16; First posted 2021-11-01 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Skin Condition
Keywords: Rice ceramide; Supplementation; Skin health
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Intervention Model Description: This will be a single arm and open-labelled prospective study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): To receive rice ceramide supplementation for 3 months
  Interventions: Dietary Supplement: Rice ceramide supplementation

INTERVENTIONS:
Dietary Supplement: Rice ceramide supplementation — At the dosage of 40mg daily for 3 months

SUMMARY:
Ceramides have been added to newer cosmetic products to improve skin barrier function and exogenously replenish skin ceramides. Of the stratum corneum intercellular lipids, Ceramides are the most effective at restoring barrier function and increasing skin hydration. Different ceramides have been incorporated into cosmetic formulations, but understanding the differences between ceramides used in formulations, or even identifying ceramides in formulations can be complex. This is mostly because of an archaic nomenclature system that is fundamentally flawed based on current scientific evidence. In the recent past, due to the unique bioactive components of rice, it has been explored to a certain limit for its components. Further, much attention has been paid to the plant ceramide with its incorporation into cosmetics and food preparations owing to its safety in contrast to animal/synthetic origin. There are reports on plant ceramide deciphering its protective effects on human skin by preventing moisture loss. It has been anticipated that ceramides, fatty acids, and cholesterol in combination with hydrocortisone (HC) can be an useful therapeutic agents against xerosis and atopic dermatitis.

The beneficial effects of oral intake of plant-derived ceramides for skin hydration and skin barrier reinforcement have been established in several studies involving animal models as well as human subjects. Ingestion of konjac ceramides has also shown positive effects in atopic dermatitis patients as well as healthy volunteers. Results showed improved skin symptoms and reduced skin allergic responses. The foregoing studies support the beneficial effects of oral intake of plant ceramides and their potential complementary and alternative therapeutic applications in the restoration and maintenance of skin barrier function. However, the findings from human study are still very limited, more detailed and comprehensive studies are still required to document the clinical efficacy of oral supplementation of ceramides. Thus, this study aims to evaluate the effects of rice ceramides consumption in improving skin health.

DETAILED DESCRIPTION:
EFFECTS OF RICE CERAMIDES IN IMPROVING SKIN HEALTH - STUDY PROTOCOL

INTRODUCTION

Background

Ceramides are important structural components of the epidermis, which plays a key role in maintaining homeostasis of the human body. Specifically, its outermost layer, known as the stratum corneum, forms a barrier between the external environment and the internal body. This barrier function serves multiple purposes including prevention of water loss and protection from foreign insult. The structure of the stratum corneum is often referred to as ''brick and mortar''. The ''bricks'' are terminally differentiated keratinocytes composed mostly of keratin filaments and filaggrin. The ''mortar'' is composed of intercellular lipids arranged into lamellar layers consisting of ceramides, free fatty acids, and cholesterol. Ceramides are the predominant lipid comprising approximately 50% of the intercellular lipid content by mass. Stratum corneum lipids are essential for maintaining skin barrier function and preventing transepidermal water loss (TEWL). Disruptions or damage to the stratum corneum can impair skin barrier function and result in TEWL.

Ceramides have been added to newer cosmetic products to improve skin barrier function and exogenously replenish skin ceramides. Of the stratum corneum intercellular lipids, Ceramides are the most effective at restoring barrier function and increasing skin hydration. Different ceramides have been incorporated into cosmetic formulations, but understanding the differences between ceramides used in formulations, or even identifying ceramides in formulations can be complex. This is mostly because of an archaic nomenclature system that is fundamentally flawed based on current scientific evidence. In the recent past, due to the unique bioactive components of rice, it has been explored to a certain limit for its components. Further, much attention has been paid to the plant ceramide with its incorporation into cosmetics and food preparations owing to its safety in contrast to animal/synthetic origin. There are reports on plant ceramide deciphering its protective effects on human skin by preventing moisture loss. It has been anticipated that ceramides, fatty acids, and cholesterol in combination with hydrocortisone (HC) can be an useful therapeutic agents against xerosis and atopic dermatitis. In addition, report also showed that topical emulsions containing ceramides possessed anti-inflammatory and skin beneficial properties. Hence, isolation of ceramide from natural source possessing anti-inflammatory and skin protective properties becomes vital.

The beneficial effects of oral intake of plant-derived ceramides for skin hydration and skin barrier reinforcement have been established in several studies involving animal models as well as human subjects. A randomized, double-blind placebo-controlled trial was conducted on women with dry skin to investigate the moisturizing effect of dietary supplement containing wheat extract enriched with ceramides and digalactosyldiglycerides (DGDG). According to the finding, there was a significant increase in skin hydration with improved associated clinical signs (itching, squamae, roughness, and redness). Ingestion of konjac ceramides has also shown positive effects in atopic dermatitis patients as well as healthy volunteers. Results showed improved skin symptoms and reduced skin allergic responses . The foregoing studies support the beneficial effects of oral intake of plant ceramides and their potential complementary and alternative therapeutic applications in the restoration and maintenance of skin barrier function. However, the findings from human study are still very limited, more detailed and comprehensive studies are still required to document the clinical efficacy of oral supplementation of ceramides. Thus, this study aims to evaluate the effects of rice ceramides consumption in improving skin health.

Objective

To determine the effects of rice ceramides consumption in improving skin health.

METHODOLOGY

Study Design

This will be an open-label, single arm, prospective interventional study that involves three-months period of rice ceramides (komercera) supplementation. Fifty subjects will be recruited via convenient sampling for this study.

Study Population

Fifty subjects are required to consume rice ceramides (komecera) supplements at the dosage of 40mg, one vegetarian capsule per day. Monthly follow-up for the duration of 3 months will be conducted to allow sufficient time for the changes to take place.

Good general healthy subjects who are free from any skin diseases, aged 20 to 45 and willing to comply with rice ceramides consumption plan will be recruited. Participant with underlying skin medical condition such as eczema, psoriasis, rosacea, atopic dermatitis, ichthyosis or vitiligo, undergoing medication plan, currently taking antimicrobial or antiviral medication, undergone major surgical procedures in the past six months, pregnant or lactating woman will be excluded from this study. All the study participants will be provided with a participant information sheet, briefly containing the research detail and a written informed consent will also be sought from each recruited participant.

Assessment will be conducted at baseline when they were first recruited, and also during their 3 times monthly follow ups. Participants will be remunerated with RM200 vouchers by the end of the study to compensate the time they spent in this research. Location of recruitment will be at public settings in Klang Valley.

Clinical Assessment

The efficacy of rice ceramides in improving the overall skin health will be assessed using the parameters below: -

* Total Wrinkle Score (TWS)
* Skin firmness and elasticity (Courage & Khazaka Cutometer®, MPA580)
* Skin hydration (Courage & Khazaka Corneometer®, CM825)
* Transepidermal Water Loss and Skin Barrier Function (Courage & Khazaka Tewameter®, TM 300)
* Skin whitening (Courage & Khazaka Mexameter®, MX18)
* Sebum Secretion (Courage & Khazaka Sebumeter®, SM815)
* Skin pH (Courage & Khazaka pH meter®, PH900)

The assessment mentioned above will be carried out using Multiprobe Adapter System (MPA), which is a non-invasive assessment.

Subjects Self-Perceived Assessment

Subject will also be required to do a self-perceived Visual Analogue Scale (VAS) to reflect their self-perceived changes.

Statistical Analysis

Demographic characteristics will be presented as categorical data, expressed in frequency and percentage. All outcomes will be analyzed as continuous dependent variables, presented as mean ± SD. The changes in clinical assessment from baseline visit to last follow-up visit will be analyzed using general linear model (GLM) for repeated measures model. Within-subjects factor will be defined as the sampling time point. Gender and age will be tested as between-subject effect. Homogeneity of the variance and covariance structure of the dependent variables will be assessed by Levene and Box M tests. Sphericity test of the residual covariance matrix will be assessed using Mauchly's sphericity test. Results will only be considered significant if P<0.05 with 95% of confidence interval. Statistical analysis will be performed using SPSS 26.0 (IBM Corp., New York, United States) for MacOS.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Free from any skin diseases
* Willing to comply with rice ceramide consumption plan
* Willing to give consent

Exclusion Criteria:

* Undergoing medication plan for skin condition
* Undergone major surgical procedures in the past six months
* Pregnant or lactating woman

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Wrinkle change | Time point 1 (month 0), time point 2 (follow-up visit month 1), time point 3 (follow-up visit month 2) and time point 4 (follow-up visit month 3)
  To be assessed using Total Wrinkle Score (TWS). TWS has a minimum value of 4 and maximum value of 20, with higher values indicating higher severity.
Change in skin firmness and elasticity | Time point 1 (month 0), time point 2 (follow-up visit month 1), time point 3 (follow-up visit month 2) and time point 4 (follow-up visit month 3)
  To be assessed using Courage & Khazaka Cutometer®, MPA580
Change in skin hydration | Time point 1 (month 0), time point 2 (follow-up visit month 1), time point 3 (follow-up visit month 2) and time point 4 (follow-up visit month 3)
  To be assessed using Courage & Khazaka Corneometer®, CM825
Change in transepidermal water loss and skin barrier function | Time point 1 (month 0), time point 2 (follow-up visit month 1), time point 3 (follow-up visit month 2) and time point 4 (follow-up visit month 3)
  To be assessed using Tewameter® TM 300
Change in skin whitening | Time point 1 (month 0), time point 2 (follow-up visit month 1), time point 3 (follow-up visit month 2) and time point 4 (follow-up visit month 3)
  To be assessed using Courage & Khazaka Mexameter®, MX18
Change in sebum secretion | Time point 1 (month 0), time point 2 (follow-up visit month 1), time point 3 (follow-up visit month 2) and time point 4 (follow-up visit month 3)
  To be assessed using Courage & Khazaka Sebumeter®, SM815
Change in skin pH | Time point 1 (month 0), time point 2 (follow-up visit month 1), time point 3 (follow-up visit month 2) and time point 4 (follow-up visit month 3)
  To be assessed using Courage & Khazaka pH meter®, PH900

SECONDARY OUTCOMES:
Adverse events | Follow-up visit month 3
  Monitor for adverse response from participants

CONTACTS AND LOCATIONS:
Overall Officials: Chung Keat Tan, PhD, Principal Investigator — UCSI University
Locations (2):
- Malaysia (2):
  - UCSI University, Cheras, Kuala Lumpur
  - Nexus Wise Sdn. Bhd., Petaling Jaya, Selangor

IPD SHARING:
Plan to Share IPD: Yes
It can be shared upon the completion of this study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anticipated to be available by the end of April 2022, for 6 months
Access Criteria: Requestor need to send in an official email to sponsor to request for the data access.

REFERENCES:
- [Background] Henderson AJ, Ollila CA, Kumar A, Borresen EC, Raina K, Agarwal R, Ryan EP. Chemopreventive properties of dietary rice bran: current status and future prospects. Adv Nutr. 2012 Sep 1;3(5):643-53. doi: 10.3945/an.112.002303. PMID 22983843
- [Background] Heule F. An oral approach to the treatment of photodamaged skin: a pilot study. J Int Med Res. 1992 Jun;20(3):273-8. doi: 10.1177/030006059202000309. PMID 1397672
- [Background] Kawano K, Umemura K. Oral intake of beet extract provides protection against skin barrier impairment in hairless mice. Phytother Res. 2013 May;27(5):775-83. doi: 10.1002/ptr.4792. Epub 2012 Sep 4. PMID 22949397
- [Background] Yeom M, Kim SH, Lee B, Han JJ, Chung GH, Choi HD, Lee H, Hahm DH. Oral administration of glucosylceramide ameliorates inflammatory dry-skin condition in chronic oxazolone-induced irritant contact dermatitis in the mouse ear. J Dermatol Sci. 2012 Aug;67(2):101-10. doi: 10.1016/j.jdermsci.2012.05.009. Epub 2012 Jun 7. PMID 22726258
- [Result] Asai S, Miyachi H. [Evaluation of skin-moisturizing effects of oral or percutaneous use of plant ceramides]. Rinsho Byori. 2007 Mar;55(3):209-15. Japanese. PMID 17441463
- [Result] Guillou S, Ghabri S, Jannot C, Gaillard E, Lamour I, Boisnic S. The moisturizing effect of a wheat extract food supplement on women's skin: a randomized, double-blind placebo-controlled trial. Int J Cosmet Sci. 2011 Apr;33(2):138-43. doi: 10.1111/j.1468-2494.2010.00600.x. PMID 20646083
- [Result] Imokawa G, Akasaki S, Hattori M, Yoshizuka N. Selective recovery of deranged water-holding properties by stratum corneum lipids. J Invest Dermatol. 1986 Dec;87(6):758-61. doi: 10.1111/1523-1747.ep12456950. PMID 3782858
- [Result] Kimata H. Improvement of atopic dermatitis and reduction of skin allergic responses by oral intake of konjac ceramide. Pediatr Dermatol. 2006 Jul-Aug;23(4):386-9. doi: 10.1111/j.1525-1470.2006.00268.x. PMID 16918640
- [Result] Miyanishi K, Shiono N, Shirai H, Dombo M, Kimata H. Reduction of transepidermal water loss by oral intake of glucosylceramides in patients with atopic eczema. Allergy. 2005 Nov;60(11):1454-5. doi: 10.1111/j.1398-9995.2005.00915.x. No abstract available. PMID 16197483